CLINICAL TRIAL: NCT06010082
Title: The Effect of Music Therapy on Psychological Status and Sleep Quality Among Pregnant Women: A Randomized Control Trail
Brief Title: The Effect of Music Therapy on Psychological Status and Sleep Quality Among Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud Khedr, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 69-D
Record Dates: First submitted 2023-08-21; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Pregnant Women
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STUDY GROUP (Experimental): Intervention group Group one (study group, 40 pregnant women): received Music Therapy intervention.
  Interventions: Behavioral: Music Therapy
- Control group (Active Comparator): Group two(the control group, 40 pregnant women):act as a control group/ waiting list
  Interventions: Behavioral: Music Therapy

INTERVENTIONS:
Behavioral: Music Therapy — Music Therapy intervention will be delivered through instructed participants to empty their bladder and then listen to music for 30 min in a semi-fowler's position with their head and shoulders raised 30° in a quiet and dim environment, listening to the music of symphonic music.

SUMMARY:
There is a strong correlation between sleep disturbance and indications of stress, anxiety, and depression. However, in Egypt no research has looked into how better sleep for expectant mothers might be achieved by inexpensive, pleasurable, non-invasive music listening. Therefore, the aim of this study was to investigate how music listening affects pregnant women's psychological status, and sleep quality.

DETAILED DESCRIPTION:
This study used a randomized controlled trial (RCT) design and adhered to the Consolidated Standards of Reporting Trials (CONSORT) guidelines. The study utilized a simple random sampling technique to select participants in proportion to the total number of pregnant women in the outpatient Medical National Institute in Damanhur city, Egypt.

ELIGIBILITY:
Inclusion Criteria:

In third trimester, 30-34th weeks of pregnancy, age ranging from 18-35 years old, singleton pregnancy, willing to participate

Exclusion Criteria:

having any physical or mental health disorders

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Depression, Anxiety, and Stress Scale | 2 months
  The Depression, Anxiety, and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety, and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content.
Sleep Quality | 2 months
  It is a standardized self-report instrument used to measure the quality and patterns of sleep during the past month. It was developed and validated by Buysse et al. in 1989. It has 9 questions. Question number 5 contains 10 sub-items (from 5a to 5j). All questions are combined to form 7 components. Scoring of answers ranged from zero to three.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No